CLINICAL TRIAL: NCT05181891
Title: Pharmaceutically-Enhanced Reinforcement for Reduced Alcohol and Smoking
Acronym: PERRAS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington State University (Other)
Responsible Party: Principal Investigator, Sterling McPherson, Professor, Washington State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18668-001
Record Dates: First submitted 2021-12-07; First posted 2022-01-06 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Alcohol Use Disorder (AUD); Nicotine Use Disorder
Keywords: Alcohol Use Disorder; Contingency Management; Incentives for Sobriety; Varenicline; Nicotine Use Disorder
MeSH Terms: conditions — Alcoholism; Tobacco Use Disorder

STUDY DESIGN:
Intervention Model Description: Phase II randomized trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (CM+TAU) Contingency Management + Treatment as Usual (Experimental): Varenicline (VC) will be supplied in .5 mg tablets once per week during the active treatment period. During the first week of treatment (Week 3) participants will be instructed to take .5 mg once per day for days 1-3, and 0.5 mg twice per day for days 4-7. The investigators will maintain a target dose of 1mg twice per day for the remaining active treatment period. Additionally, participants will also receive Take Control counseling via video. Participants in CM+TAU will receive reinforcement for submitting urine samples that test negative for recent alcohol use.
  Interventions: Behavioral: Contingency Management
- (NC+TAU) No Contingency + Treatment as Usual (Active Comparator): Varenicline (VC) will be supplied in .5 mg tablets once per week during the active treatment period. During the first week of treatment (Week 3) participants will be instructed to take .5 mg once per day for days 1-3, and 0.5 mg twice per day for days 4-7. The investigators will maintain a target dose of 1mg twice per day for the remaining active treatment period. Additionally, participants will also receive Take Control counseling via video. NC+TAU will receive reinforcement for submitting any urine sample, regardless of test results.
  Interventions: Behavioral: Non-contingent control

INTERVENTIONS:
Behavioral: Contingency Management — Incentives for submitting negative-alcohol urine samples
  Arms: (CM+TAU) Contingency Management + Treatment as Usual
Behavioral: Non-contingent control — Incentives for submitting urine samples
  Arms: (NC+TAU) No Contingency + Treatment as Usual

SUMMARY:
Using a randomized controlled trial (RCT), the goal of this study is to evaluate the ability of evidence based behavioral treatment (contingency management: CM) to significantly decrease alcohol use and cigarette smoking among treatment-seeking smokers with an alcohol use disorder (AUD) who have initiated pharmacotherapy (varenicline; VC) for smoking cessation.

DETAILED DESCRIPTION:
This randomized, placebo-controlled trial to determine the effectiveness of contingency management for reducing alcohol use and cigarette smoking among adults who want to quit or reduce their co-addiction. Contingency management is a powerful and cost-effective technique that has been used successfully for decades to promote abstinence from benzodiazepines, cocaine, tobacco, etc. Contingency management, and a non-contingent control condition will be used combined with varenicline (VC) and manualized counseling in the form of module videos.

ELIGIBILITY:
Inclusion Criteria:

1. 4 or more standard drinks on the same occasion for women (5 or more standard drinks on the same occasion for men) on at least 4 occasions in the prior 30 days
2. Seeking AUD treatment
3. Seeking smoking cessation treatment
4. Aged 18+ years
5. DSM-5 diagnosis of AUD
6. Currently smoking daily according to PhenX Smoking Status (100 or more lifetime cigarettes plus current daily smoking)
7. Ability to read and speak English
8. Ability to provide written informed consent
9. Breath alcohol of 0.00 during informed consent
10. Provision of at least 1 EtG-positive urine test at any time during the induction period and at least one COT-positive urine test at any time during the induction period; and
11. Attended at least 4 of 6 possible visits during the induction period.

Exclusion Criteria:

1. Significant risk of dangerous alcohol withdrawal, defined as a history of alcohol detoxification or seizure in the last 12 months and expression of concern by the participant about dangerous withdrawal
2. Currently receiving any pharmacotherapy for alcohol
3. Currently receiving any pharmacotherapy for smoking
4. No suicide attempt in the last 20 years and
5. Any other medical (discernable by initial blood tests) or psychiatric condition that Drs. Layton or Rodin determine would compromise safe participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 205 (Estimated)
Dates: Start 2022-07-11 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in Biochemically Verified Alcohol Use | 12-week treatment period and 7-month follow-up period
  Consumption of alcohol between participants randomized to CM+TAU vs NC+TAU assessed by alcohol EtG values (collected 3x weekly from weeks 1-14, and once at weeks 18, 30, 42).
Change in Biochemically Verified Tobacco Use | 12-week treatment period and 7-month follow-up period
  Consumption of tobacco between participants randomized to CM+TAU vs NC+TAU assessed by tobacco CO and COT values (collected 3x weekly from weeks 1-14, and once at weeks 18, 30, 42).

SECONDARY OUTCOMES:
Change in Self Reported Alcohol Use | 12-week treatment period and 7-month follow-up period
  Consumption of alcohol between participants randomized to CM+TAU vs NC+TAU assessed by participant self report (collected 3x weekly from weeks 1-14, and once at weeks 18, 30, 42).
Change in Self Reported Tobacco Use | 12-week treatment period and 7-month follow-up period
  Consumption of tobacco between participants randomized to CM+TAU vs NC+TAU assessed by participant self report (collected 3x weekly from weeks 1-14, and once at weeks 18, 30, 42).

CONTACTS AND LOCATIONS:
Overall Officials: Sterling M McPherson, PhD, Principal Investigator — Washington State University
Locations (1):
- Washington State University, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No